CLINICAL TRIAL: NCT05186519
Title: Amputation Associated Factors and Prediction Model in Diabetic Foot Patients : A Retrospective Cohort Study
Brief Title: Amputation Associated Factors and Prediction Model in Diabetic Foot Patients
Status: Completed | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CT2021-10-22
Record Dates: First submitted 2021-12-09; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Diabetic Foot
Keywords: Diabetic Foot; Amputation; Cohort Study; Predict model
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetic foot can lead to adverse consequences such as amputation and death, which seriously endangering the physical and mental health and quality of life for patients.

The aim of this study is to assess factors associated with the occurrence of amputation events in the diabetic foot patients based on a retrospective cohort and to construct a prediction model for patients at high amputated risk.

DETAILED DESCRIPTION:
Diabetic foot is one of the major complications observed in patients with diabetes. Diabetic foot can lead to non-traumatic lower-limb amputation (LLA), and is confirmed to be associated with cognitive decline and worsening quality of life. Previous studies indicated that diabetics had a 25% lifetime risk of developing diabetic foot, and 14% to 24% of those require amputation. In patients with poor results of conservative treatment, amputation is the main terminal treatment option to avoid the spread of infection.

Amputation in diabetic foot patients may linked to different causes, including inflammatory, infectious and malignant conditions. A retrospective cohort based on Shandong Provincial Qianfoshan Hospital Healthcare Big Data Platform is conducted to evaluate the progression and prognosis of diabetic foot patients. A prediction model will be developed to identify high-risk diabetic foot patients of amputation and provide a scientific basis for personalized clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetic foot
* Hospitalized patients
* No history of amputation

Exclusion Criteria:

* Patients with Bone Neoplasms
* Patients with osteomyelitis not caused by diabetes
* Patients with amputation caused by severe peripheral vascular disease not caused by diabetes
* Traumatic Amputations
* Patients in shock on admission
* Patients discharged against medical advice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic foot who were hospitalized in The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital between January 1, 2015 and October 15, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
All non-traumatic amputate events | through study completion, an average of 2.2 year
  The main outcome was any non-traumatic amputation events among patients with diabetic foots including removing all of a limb or extremity (major amputation) or a portion of a limb or extremity (minor amputation).

SECONDARY OUTCOMES:
Composite outcomes of serious adverse | through study completion, an average of 2.2 year
  Including amputations, deaths and other adverse outcomes
All-cause mortality | through study completion, an average of 2.2 year
  All-cause mortality during hospitalization in patients with diabetic foot.
Length of stay in hospital | through study completion, an average of 2.2 year
  Hospital length of stay for diabetic foot treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yibing, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided